CLINICAL TRIAL: NCT02138604
Title: Non Invasive dP/dt is Not a Good Index to Detect an Acute Ischemic Myocardial Dysfunction in Emergency Department (ED)
Brief Title: Non Invasive dP/dt to Detect an Acute Ischemic Myocardial Dysfunction in Emergency Department
Acronym: dP/dtAMDED
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Non invasive dP/dt is not a good index to detect an acute ischemic myocardial dysfunction in emergency department (ED), University of Monastir
Other Study IDs: dp/dt to detect AMD in ED
Record Dates: First submitted 2014-04-08; First posted 2014-05-14 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Acute Myocardial Ischemia
Keywords: chest pain; myocardial ischemia; acute myocardial dysfunction; plethesmography; non invasive dP/dt
MeSH Terms: conditions — Chest Pain; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Most patients presenting to the emergency department with chest discomfort have a nonischemic ECG and biomarkers of myocardial necrosis within normal limits. These patients are routinely admitted to hospital because of diagnostic uncertainty for occult MI or ischaemia.

Acute myocardial ischemia is associated with acute mycardial dysfunction We tested a non-invasive plethysmographic arterial pressure change index of myocardial performance (dP/dt) that could be added to the diagnostic triage of ischaemia in the ER avoiding unnecessary admissions.

DETAILED DESCRIPTION:
For patients with chest pain , the ECG remains the most important initial risk assessment tool. Myocardial ischemia or infarction is highly likely in patients with significant ST segment changes on the ECG or elevation in myocardial markers of necrosis. Identification of high-risk patients is more difficult in those with non ischemic ECG and negative markers on presentation.

One of the most sensitive indices of contractility is the rate of increase of intraventricular pressure during isovolumetric contraction, (left ventricular dP/dt and arterial dP/dt). Dp/dt (dP/dt ejc ) represents the rate of change of pressure during ejection. It has been shown that cardiac contractility and dP/dt decreases during acute myocardial ischemia.

We theorized that a higher value of dP/dt would be found for non ischemic chest pain than during ischemic chest pain because ischemia reduces myocardial contractility, whereas chest pain of non cardiac origin increases dP/dt by the stress of the pain itself.

The current study describes a noninvasive plethysmographic dP/dt changes in patients presenting at the emergency department with acute chest pain, which could be added to the diagnostic triage of ischemia in the ED, thus decreasing the number of unnecessary admissions.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 year old
* Chest pain that lasted less than 12 hours

Exclusion Criteria:

* traumatic chest pain
* arrythmias
* STEMI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department with acute chest pain
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
plethysmographic dP/dt cardiac output value in patients with acute chest pain | at admission
  compare the noninvasive dP/dt values in the two study groups: Acute Coronary syndrome (ACS) and non ACS.
  the diagnostic of ischemic origin of chest pain is based on anamnestic, electrocardiographic, and necrosis enzymes.

CONTACTS AND LOCATIONS:
Overall Officials: semir Nouira, Pr, Principal Investigator — University of Monastir
Locations (1):
- Nouira Semir, Monastir, CHU Fattouma Bourguiba, Tunisia

IPD SHARING:
Plan to Share IPD: No